CLINICAL TRIAL: NCT01408433
Title: Single Embryo Transfer of a Euploid Embryo Versus Double Embryo Transfer: A Randomized Controlled Trial
Brief Title: Single Embryo Transfer of a Euploid Embryo Versus Double Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RMA-2011-01
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: embryo transfer; in-vitro fertilization (IVF); pre-implantation diagnosis (PGD); infertility; single embryo transfer; two embryo transfer; double embryo transfer
MeSH Terms: conditions — Infertility | interventions — Single Embryo Transfer; Fertilization in Vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Embryo Transfer (Other): Patients will have a single, chromosomally normal embryo transferred.
  Interventions: Other: Single Embryo Transfer
- Double Embryo Transfer (Other): Patients will have two (2) untested embryos transferred.
  Interventions: Other: Double embryo transfer

INTERVENTIONS:
Other: Single Embryo Transfer — single embryo transfer of a chromosomally normal embryo
  Other Names: pre-implantation genetic diagnosis (PGD); in-vitro fertilization (IVF)
  Arms: Single Embryo Transfer
Other: Double embryo transfer — two (2) embryo transfer of untested embryos
  Other Names: two embryo transfer; in-vitro fertilization (IVF)
  Arms: Double Embryo Transfer

SUMMARY:
This study seeks to compare the pregnancy and delivery rates of patients who undergo a single embryo transfer, when the embryo has been tested and determined to be chromosomally normal, with pregnancy and delivery rates of patients who undergo a two (2) embryo transfer of untested embryos.

DETAILED DESCRIPTION:
This study will recruit patients from the NJ/NY/CT/eastern PA area only.

Twin and higher-order multiple pregnancies are the most common and most significant complication of pregnancies conceived through assisted reproductive technologies (ART). Twin rates in in vitro fertilization (IVF) cycles are approximately 30%. These pregnancies have increased complications for both the mother and the babies. A singleton, one baby, is the safest outcome for an IVF cycle. The surest way to reduce the risk of multiple births in IVF cycles is to transfer fewer embryos. Prior studies on single embryo transfer (SET) have shown decreased pregnancy rates because of the difficulty in selecting which embryo to transfer. Being chromosomally normal is necessary for the delivery of a healthy baby. The investigators are now able to screen all 24 chromosomes of an embryo with greater than 97% accuracy within four hours, allowing for a fresh embryo transfer of a tested embryo, using Comprehensive Chromosome Screening (CCS). This study seeks to show that the transfer of a single CCS-normal embryo will result in delivery rates equal to those resulting from a two embryo transfer, the current standard of care in IVF.

Patients will undergo IVF according to the protocol recommended by their primary doctor. On the day of egg retrieval, all mature eggs will be fertilized by intracytoplasmic sperm injection (ICSI) per routine laboratory protocol. Embryos will then be cultured out to day 5 per routine laboratory procedure. The embryos will be assessed by the embryologist on day 5 to determine if the patient is a candidate for a fresh transfer. Patients who are a candidate for fresh transfer will be randomized into either the single embryo transfer of a chromosomally normal embryo group or the double, untested embryo group. Patients will have a 50:50 chance of being in the single or double embryo transfer group. Embryos in the single embryo group will undergo biopsy for CCS and patients will then undergo transfer of the morphologically best, chromosomally normal embryo. Additional embryos will be cryopreserved. Patients in the double embryo transfer group will undergo a two embryo transfer. Additional embryos will be cryopreserved. If patients are not a candidate for a fresh transfer (potentially because of endometrial lining development, risk of ovarian hyperstimulation syndrome, or embryos that are not suitable for biopsy on day 5), they will still be randomized into either the single or double embryo transfer group. Patients in the single embryo transfer group will have all embryos biopsied for CCS prior to being frozen. Patients will then immediately undergo a synthetic frozen embryo transfer cycle in accordance with their randomization. Patients in the double embryo transfer group will have their embryos frozen and will then immediately prepare for a synthetic frozen embryo transfer cycle in accordance with their randomization. Any patient who does not become pregnant during their fresh transfer cycle will immediately undergo a synthetic frozen embryo transfer cycle in accordance with their original randomization.

All clinical follow up will be per routine regarding pregnancy testing, early pregnancy monitoring and subsequent transfer of care to the patient's obstetrician. If clinical miscarriage occurs, cells from the products of conception will be collected, if possible, and submitted for genetic analysis. If the pregnancy progresses to delivery, a buccal swab (small swab touched to the inside of the baby's cheek) will be collected and submitted for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Maximum of one (1) prior failed IVF cycle (a failed cycle is any cycle that did not deliver. Pregnancy losses are failed cycles. Ok to participate as a recipient in an egg donor cycle.)
2. Female partner less than 43 years old at time of onset of IVF cycle
3. Maximum prior day 3 follicle stimulation hormone (FSH) level of 12 (in RMA NJ laboratory)
4. Minimum anti-mullerian hormone (AMH)of 1.2 within 1 year
5. Normal uterine cavity demonstrated by saline sonogram, hysterosalpingogram or hysteroscopy within 1 year.
6. Male partner with greater than 100,000 total motile spermatozoa. Donor sperm ok.
7. Body Mass Index (BMI) less than or equal to 30 kg/m2.

Exclusion Criteria:

1. Diagnosis of chronic anovulation (cycles typically longer than 90 days)
2. Diagnosis of endometrial insufficiency- prior cycle with endometrial thickness less than 6mm, abnormal endometrial echotexture, persistent endometrial fluid.
3. Clinical indication of aneuploidy screening (i.e. history of loss of chromosomally abnormal pregnancies)
4. Clinical indication for PGD for single-gene disorder (i.e. PGD is needed to select against the transfer of embryos affected with a specific condition)
5. Use of testicular aspiration or biopsy procedures to obtain sperm
6. Unevaluated ovarian mass or surgically confirmed stage IV endometriosis
7. Presence of hydrosalpinges which communicate with the endometrial cavity
8. Any contraindication to undergoing in vitro fertilization

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Live birth rate per randomized patient (single embryo transfer vs. 2 embryo transfer) | 2 years
  Compare live birth rates of patients who have a single embryo transfer of a chromosomally normal embryo with the live birth rates of patients who have two, untested embyros transferred.

SECONDARY OUTCOMES:
Twin live birth rate | 2 years
  Compare twin live birth rates of patients who have a single embryo transfer of a chromosomally normal embryo with the twin live birth rates of patients who have two, untested embryos transferred.
Sustained implantation rate (number of viable fetuses beyond the first trimester per embryo transferred) | 2 years
  Compare sustained implantation rates of patients who have a single embryo transfer of a chromosomally normal embryo with the sustained implantation rates of patients who have two, untested embryos transferred.
Live birth rate per embryo transfer | 2 years
  Compare live birth rates per transfer of patients who have a single embryo transfer of a chromosomally normal embryo with the live birth rates per transfer of patients who have two, untested embryos transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — RMA NJ
Locations (2):
- United States (2):
  - Reproductive Medicine Associated of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Associated of Pennsylvania at lehigh Valley, Allentown, Pennsylvania

REFERENCES:
- [Derived] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942